CLINICAL TRIAL: NCT05513040
Title: Clinical Course of Functional Dyspepsia and Factors Predicting Outcome in Patients Receiving Medication-based Treatment
Status: Recruiting | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Other Study IDs: KY20222180-F-3
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional dyspepsia (FD) is one of most common chronic gastrointestinal disorders. Several types of drugs were demonstrated to be effective in reduction or remission of symptoms and severity of FD, including proton pump inhibitors (PPI), Tricyclic antidepressant and prokinetics. However, the clinical course of FD after taking medication-based treatment was unknown. Furthermore, 20-50% patients remained persistent or worsening of dyspepsia symptoms after treatment. Previous studies have suggested psychological factors (eg. anxiety, sleep disturbance) were related to less improvement of symptoms in natural clinical course. However, there is limited evidence in terms of clinical and psychological factors for less improvement in patients receiving medication treatment for dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years old
2. Patients who met Rome IV criteria
3. Normal upper endoscopy and abdominal ultrasonography within one year

Exclusion Criteria:

1. Patients with local or systemic diseases which may cause dyspeptic symptoms:

   Known active peptic ulcer, cholecystitis, gallstone, gastrointestinal obstruction, gastroparesis, and etc.; Known acute or chronic injury of liver or kidney; Obvious hematological abnormality, or endocrine and metabolic diseases; Known malignancy; Obvious cardiovascular or cerebrovascular diseases (such as coronary heart disease, arrhythmia, cerebral infarction and etc.; Other conditions which may be associated with dyspeptic symptoms (such as NSAIDs associated dyspepsia)
2. organ failure defined by Marshall standard
3. severe psychiatric illnesses
4. known malignancy
5. pregnancy or lactation
6. unable to provide consent
7. suspected or identified bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years old who met criteria of functional dyspepsia defined by Rome IV were eligible for our study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
score of 4 (slightly better) or 5 (much better) on a 5-point Likert scale assessing symptom improvement at 6 months after the initial visit | 6 months
  A 5-point likert scale was used for accessing symptom relief. 1. Worse, 2,slightly worse, 3.same, 4.slightly better, 5.much better. A score of 4 or 5 was classified as relief response.

SECONDARY OUTCOMES:
subtypes of functional dyspepsia | 6 months
  functional dyspepsia was classified into three subgroups：(1) Postprandial Distress Syndrome, defined as Bothersome postprandial fullness or/and Bothersome early satiation. (2) Bothersome epigastric pain AND/OR Bothersome epigastric burning. (3) mixed syndrome, defined when postprandial distress syndrome and epigastric pain syndrome presented simultaneously.
Short Form of Nepean Dyspepsia Index (SF-NDI) | 1 day
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hospital anxiety and depression scale | 1 day
  Anxiety and depression of patients are assessed by using Hospital Anxiety and Depression Scale.It contains 14 items (7 anxiety and 7 depression), which assess symptoms experienced during the past week on a 0-3 scale. A subscore of > 8 for depression or anxiety would indicate a clinical case.
Quality of Life scores assessed by Patient-reported outcomes measurement information system (PROMIS) Global-10 questionaire. | 1 day
  Quality of Life scores assessed by Patient-reported outcomes measurement information system (PROMIS) Global-10 questionnaire. PROMIS Global-10 is a newly validated 10-question survey used to assess health care-related quality of life measures for the general population.
  It's a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient and a better quality of life.
the change of Global Overall Symptom score (GOSS) | 1month, 3 months, 6 months,12 months
  The GOSS consists of 10 cardinal items (epigastric pain, epigastric discomfort, Heartburn, acid regurgitation, upper abdominal bloating, belching, nausea, early satiety, postprandial fullness, other epigastric symptoms(eg. epigastric burning). Each item can be scored from 1 (no) to 7 (worst).
Adequate relief rate | 1month, 3 months, 6 months,12 months
  Patients had adequate relief of symptoms in the past 7 days.
the change of Functional dyspepsia symptom diary (FDSD) score | 1month, 3 months, 6 months,12 months
  The FDSD consists of 5 cardinal items (burning in the stomach, stomach pain, bloating, postprandial fullness, and early satiety) and 3 supplementary items (nausea, burping/belching rating, and burping/belching bother). Each item can be scored from 0 (no) to 10 (worst).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing 986 Hospita, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi